CLINICAL TRIAL: NCT07031128
Title: Evaluating the Impact of Alpha Ketoglutarate (AKG), a Geroprotector, in Reducing Morbidity and Improving Patient-Centred Outcomes After Coronary Artery Bypass Grafting Surgery in Resilient and Poorly-Resilient Patients: A Double-Blind Placebo-Controlled Clinical Trial
Brief Title: Alpha Ketoglutarate Enhances Geroprotection In Surgery (AEGIS)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Wellcome Leap Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023/00747
Record Dates: First submitted 2024-10-16; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-09

CONDITIONS: CABG
Keywords: Geroprotector; Alpha-ketoglutarate
MeSH Terms: interventions — Ketoglutaric Acids

STUDY DESIGN:
Intervention Model Description: Recruited patients will be randomized 1:1 to either receive AKG or placebo, stratified to each institution. Following successful randomization, each patient will be assigned a unique patient study number and a unique medication kit number.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AKG (Experimental): To receive AKG tablets (1g a day, once a day, taken orally)
  Interventions: Dietary Supplement: Alpha-ketoglutarate
- Placebo (Placebo Comparator): To receive placebo tablets (1g a day, once a day, taken orally)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha-ketoglutarate — Alpha-ketoglutarate supplements
  Arms: AKG
Dietary Supplement: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
One of the most common major surgeries that older patients undergo is coronary artery bypass grafting surgery (CABG), which is performed in approximately 400,000 patients in the United States each year. CABG invokes a massive surgical stress response, with systemic epinephrine increasing 33-fold and norepinephrine increasing 3-fold. Initially, local tissue injury results in a sterile inflammation, releasing damage-associated molecular patterns (DAMPS). DAMPS activate neutrophils, bringing a cascade of cytokines, complement, and coagulation changes. Activation of nociceptors results in a neurometabolic response involving the sympathetic nervous system and hypothalamus-pituitary axis. This brings about systemic effects including changes in basal metabolic rate, hyperglycemia, lipolysis, negative nitrogen balance, and release of cytokines and complement. Although the surgical stress response is essential for wound healing and is usually self-limiting, an exaggerated response may occur resulting in multiple organ dysfunction.

The acute phase of the surgical stress response is often followed by secondary insults that may be either sterile or pathogen-induced (such as postoperative infection).In the "two-hit" model of surgical stress response, there is an exaggerated response even to minor insults in vulnerable individuals who were primed by the initial stress response. Changes in the microbiome may also occur, developing a "pathobiome" that may enter the systemic circulation. If left unchecked, this second hit may result in the development of systemic inflammatory response syndrome (SIRS) and multi-organ failure.

Chronological ageing changes the innate and adaptive immunity of patients. Biological hallmarks of aging such as genomic instability, mitochondrial damage, glycation of proteins, and cellular senescence all result in increased oxidative stress and systemic inflammation. Aging brings about a pro-inflammatory innate immune responsiveness that often occurs even in the absence of an inflammatory threat. This is termed inflammaging. Paradoxically, inflammaging is associated with an increased risk of infection and poor response to stressful events. At the same time, there is an age-associated loss of T-cell function, particularly in naïve CD8 T-cells. This deficit is termed immunosenescence and is characterised by reduced pathogen recognition, chemotaxis, and phagocytosis.

DETAILED DESCRIPTION:
Within 24 hours of surgery, single-cell mass cytometry identified signalling changes in immune cell subsets that characterise the phenotypic and functional immune response to surgery. These signals accounted for 40-60% of observed patient variability, and strong correlations were found between these immune signatures with the speed of recovery from fatigue, pain, and functional impairment. In another study, Fragiadakis found that the preoperative immune state was also predictive of recovery from surgery, with toll-like receptor (TLR) 4 signalling in cluster of differentiation (CD) 14+ monocytes accounting for 50% of observed variance in clinical recovery. Furthermore, the group showed that patients undergoing an intermediate risk cardiac surgery had a significantly higher risk of developing multi-organ failure when their cytokine response profile was highly proinflammatory after stimulation with Escherichia coli-derived lipopolysaccharide . Another study showed that patients' immune response after surgery and immune profile before surgery predicted the development of surgical site complications in abdominal surgery. Taken together, these studies were consistent in suggesting that immune profiles play a major role in surgical resilience.

Therefore, it is postulated that giving a geroprotector in the perioperative period can mitigate the aging-related immune changes and prevent a dysfunctional surgical stress response, directly impacting surgical resilience. AKG is a geroprotector that benefits patients undergoing cardiac surgery. Plasma concentrations of AKG are reduced in patients with ischemic heart disease and it is possible that this aggravates myocardial ischemic injury during CABG. AKG supplementation during cardiopulmonary bypass significantly decreased ischaemic injury markers (creatine kinase MB and troponin T) by 30-50% in patients undergoing heart surgery, secondary to improved myocardial oxygen extraction.

AKG has beneficial effects beyond its cardiac effects. AKG is an intermediate in the Krebs cycle which is involved in various metabolic and cellular pathways as a signalling molecule, energy source, and precursor of amino acid synthesis. AKG is an anti-oxidative agent and a significant source of cellular adenosine triphosphate (ATP). Therefore, AKG plays an important role in multiple metabolic processes, and has been shown to preserve skeletal muscle, improve renal function, and protect neurological function. AKG is also a regulator of cell signalling pathways that maintain energy homeostasis, including mechanistic target of rapamycin (mTOR) and AMP-activated protein kinase (AMPK). By reducing the triggers of oxidative stress and hypoxia, AKG can moderate inflammation. AKG also has immune-modulatory properties. It modulates monocyte and neutrophil function by increasing phagocytosis and reactive oxygen species (ROS) intermediate production, macrophages by enhancing cytokine production, and lymphocytes by enhancing their proliferation.

Hypothesis Inflammaging and immunosenescence renders the older patient vulnerable to a dysfunctional surgical stress response.

ELIGIBILITY:
Inclusion Criteria

1. Scheduled for elective CABG with cardiopulmonary bypass
2. Aged 50 years and above
3. Adequate cognitive function to be able to give informed consent

Exclusion Criteria

1. Patients already taking AKG as a supplement
2. Substance abuse disorder either untreated or treated
3. Post-traumatic stress disorder, bipolar disorder, Schizophrenia, or any other untreated or poorly controlled mental health or mood disorder, or history of hospitalization due to mental health condition in the past 3 years, cognitively impaired patients
4. HIV/AIDS
5. Patients undergoing or scheduled to undergo chemotherapy or any other treatment for malignancy
6. Patients scheduled for immunosuppressant therapy for transplant
7. Patients with an active infection requiring antibiotic or antiviral therapy
8. Pregnant women / planning to conceive / breastfeeding women
9. Patients who are taking chronic anti-inflammatory drugs e.g., NSAIDS
10. Patients who are hypersensitivity to AKG or placebo or any components of the respective tablets to be administered

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite of systemic inflammatory response syndrome (SIRS) and at least 1 organ system | Postoperative till day 90
  The primary outcome will be a composite of systemic inflammatory response syndrome (SIRS) and at least 1 organ system dysfunction in the systems below.
  * SIRS; and
  * Cardiovascular dysfunction; and/or
  * Neurologic dysfunction; and or
  * Renal dysfunction; and/or
  * Respiratory dysfunction; and or
  * Coagulation dysfunction

SECONDARY OUTCOMES:
Other Clinical Outcomes which may be impacted by AKG - Muscle Mass | Postoperative till day 90
  * Circumferential measurements of arms and calves in cm
  * Triceps fold thickness in cm
Other Clinical Outcomes which may be impacted by AKG - Muscle Strength | Postoperative till day 90
  • Hand grip strength in kg
Other Clinical Outcomes which may be impacted by AKG - Infections Acquired | Postoperative till day 90
  * Surgical site infection: observational & charting review
  * Hospital-acquired infection: observational & charting review
Other Clinical Outcomes which may be impacted by AKG - Long-term Outcomes | Postoperative till day 90
  * Inflammation
  * Cardiac
  * Neurological
  * Renal
  Long-term Outcomes will be determined by charting reviews to determine if there are failure of the above listed organ systems
Other Clinical Outcomes which may be impacted by AKG - Mortality | Postoperative till day 90
  • Mortality from any cause
  To be determined by charting reviews and observation
Resource Utilization - Length of stay | Postoperative till day 90
  * ICU length of stay (days)
  * Hospital length of stay (days)
  To be determined by charting reviews and observation
Resource Utilization - Discharge | Postoperative till day 90
  • Patient discharge location
  To be determined by charting reviews
Resource Utilization - Unplanned readmission | Postoperative till day 90
  • Unplanning readmission from any cause
  To be determined by charting reviews
Resource Utilization - Hospital bill size | Postoperative till day 90
  • Cost of hospital stay (SGD) To be determined by charting reviews and requesting bill information from participants
Biological Ageing - Methylation & Dynamic Clocks | Postoperative till day 90
  Various computer algorithms will be used to determine DNA methylation status
Identification of Immune or Inflammatory Markers | Postoperative till day 90
  Blood samples will be collected and laboratory tests will be conducted to identify immune and inflammatory biomarkers.
  Known inflammatory biomarkers such as CRP, IL-6, TNF-α,IL-1α,IL-10 and IL-8 (not exhaustive) and newly identified biomarkers will be investigated to look at how CABG surgery changes a patient's frailty status and whether AKG has an impact on these biomarkers.
Investigations on Immune Reactivity's Relation with Surgical Resilience | Postoperative till day 90
  • To systematically address the endogenous signalling pathways conferring resilience of immune cells from patients with and without AKG treatments, peripheral blood mononuclear cells (PBMCs) will be stimulated with a panel of agonists that activate different toll-like receptors. Multiplexed cytokine analysis will be conducted on stimulated and control PBMCs. High dimensional, subset-specific, flow cytometry will be utilized at all points to assess changes in surface markers that indicate immune activation, immune regulation and senescence/exhaustion.
Patient-Centred Outcomes - Frailty | Postoperative till day 90
  The study team will determine the patient's frailty based on observation, charting reviews and available clinical information.
Patient-Centred Outcomes - Pain | Postoperative till day 90
  • Self-reported pain scores at rest and on movement using visual analogue scale (0 - 10)
Patient-Centred Outcomes - Disability | Postoperative till day 90
  Study team will determine the patient's diability status base on observation. This will be conducted pre- and post- operation to determine if there is any changes in disability status due to operation, and if and how AKG has impacted this status.
Patient-Centred Outcomes - Quality of Life | Postoperative till day 90
  • EuroQol 5 Dimension (EQ-5D)
Patient-Centred Outcomes - Fatigue | Postoperative till day 90
  • FACIT (Functional Assessment Of Chronic Illness Therapy)
Patient-Centred Outcomes - Depression | Postoperative till day 90
  • Hospital Anxiety and Depression Scale (HADS)
Patient-Centred Outcomes - Patient Satisfaction | Postoperative till day 90
  • Patient satisfaction score using visual analogue scale (0 - 10)

OTHER OUTCOMES:
Changes in Immune Status | Postoperative till day 90
  Comparison between study groups for changes, if any, in gene expression levels using peripheral blood transcriptomics
Changes in Gut Microbiome | Postoperative till day 90
  Comparison between study groups for changes, if any, in gut microbiome via shotgun sequencing to identify microbiome population pre-AKG, pre-op and post-op.
Impact of AKG on Cardiometabolic Status | Postoperative till day 90
  Comparison between study group for changes in cardiometabolic status using metabolic profiling to elucidate the pathway(s) of AKG and ischemic cardio protection.
Investigations into Immune Dysregulation and Inflammation | Postoperative till day 90
  Multiomics platform will be used to identify underlying pathways involved in immune dysregulation and inflammation, if any, and how these pathways are affected by the consumption of AKG pre- and post- operation.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Kah Ti, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No